CLINICAL TRIAL: NCT05224232
Title: Access Socket Protocol: Evaluation of Comfort and Quality of Life Associated With the Use of a Soft Socket for Femoral Prosthesis
Brief Title: Protocole Access-Socket
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Collaborators: Institution Nationale des Invalides (Other); Hôpital d'Instruction des armées Percy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRR-CLP-2020-9
Record Dates: First submitted 2022-01-03; First posted 2022-02-04 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Lower Limb Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access Socket (Experimental): Patients will be fitted with the access socket
  Interventions: Device: Access Socket
- Rigid socket (Active Comparator): Patients will be fitted with their usual rigid socket
  Interventions: Device: Rigid socket

INTERVENTIONS:
Device: Access Socket — During a period of 4 weeks, patients will live in their usual environment with the soft socket (Access-Socket)
  Arms: Access Socket
Device: Rigid socket — During a period of 4 weeks, patients will live in their usual environment with their usual rigid socket
  Arms: Rigid socket

SUMMARY:
Lower limb amputation has a definitive impact on a person's locomotor abilities, considerably reducing his or her autonomy in everyday life. 50% of lower limb amputees in France are trans-femoral. The femoral prosthesis must be adapted to allow the amputee to walk in everyday situations and to make the range of activities practiced by non-amputees accessible to them. Sitting posture, which represents an important part of a day, must also be comfortable.

Comfort will be closely linked to the socket, which ensures the transmission of the mechanical actions of the prosthesis to the body of the amputee through the residual limb. This must be done without damaging the integrity of the biological tissues at the interface. The challenge is therefore to transmit the mechanical actions inherent to the use of the prosthesis while being as comfortable as possible. The most common form of femoral socket is the one with included ishions, which by its structure limits the rotation of the socket around the residual limb. However, it limits hip joint amplitudes, which significantly impacts comfort during walking, especially when the individual must evolve in constraining environments (irregular terrain, slopes, uphill, downhill). Comfort is also limited when putting the prosthesis in place and when sitting, because of the limits of the socket that go up into the groin and the buttock. Discomfort can also be induced by contact and clamping surfaces.

Only 42% of amputees are satisfied with their sockets. An uncomfortable or wound-inducing brace will not be worn or will be worn only a little, which can increase the risk of comorbidities. One solution to the comfort issue could be the Access Socket (AS) soft socket, which is exactly the same shape and manufacturing principles as the Rigid Included Carbon Socket (ER), but combines a rigid structure with soft areas. These soft areas allow pressure to be distributed within the socket, allowing for some deformation, while maintaining the mechanical properties necessary for walking.

The objective of this study is to compare the comfort perceived by amputees when wearing an AS soft socket versus their RE, both sockets being mounted identically on the patients' usual medical devices.

The hypothesize is that scores on the various comfort, satisfaction, and mobility scales should be better when patients wear the soft socket compared to the rigid socket.

In this multicenter, randomized, cross-over study, patients will wear the rigid socket and then the access-socket (or vice versa), over a 4-week period for each socket. The two sockets will have an identical shape and will be mounted in the same way on the patients' medical device. At the end of each 4-week period, patients will fill out self-questionnaires (PEQ, SCS, PLUS-M, ESAT and SF-36) to evaluate their comfort, satisfaction and ambulation.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral trans-femoral amputees;
* Fitted with a rigid carbon insert;
* Any type of stump;
* Any etiology;
* Person able to understand simple commands, to read, write and give informed consent or having the possibility to be accompanied by a trusted person in case of inability to write or read independently;
* Person who has given informed consent;
* Person who has reached the age of 18 years;
* Person affiliated to the french social security system

Exclusion Criteria:

* Fitted with a collar fixed on a socket
* Using SHA for inserting the insert;
* Pregnant or nursing woman;
* Minor;
* Person of full age under legal protection or unable to give consent;
* Person under guardianship or curatorship;
* Person under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Comfort | Comfort will be evaluated after 4 weeks of wearing the rigid socket and after 4 weeks of wearing the Access-Socket
  Score of the Utility subscale of the Prosthesis Evaluation Questionnaire. The score ranges from 0 to 10. A higher score mean a better outcome.

SECONDARY OUTCOMES:
Satisfaction with the socket | Satisfaction will be evaluated after 4 weeks of wearing the rigid socket and after 4 weeks of wearing the Access-Socket
  Score of the french version of the Quebec USer Evaluation of Satisfaction With Assistive Technology. The score ranges from 0 to 5. A higher score mean a better outcome.
Quality of lie | Qualitify of life will be evaluated after 4 weeks of wearing the rigid socket and after 4 weeks of wearing the Access-Socket
  Score of the Short-Form 36 questionnaire. The score ranges from 0 to 100. A higher score mean a better outcome.
Mobility | Mobility will be evaluated after 4 weeks of wearing the rigid socket and after 4 weeks of wearing the Access-Socket
  Score of the Mobility subscale of the PLUS-Mobility questionnaire. This scale needs to convert a raw score (from 12 to 60) in a T-score (from 21.8 to 71.4). A higher score means a better outcome
Comfort during specific situation | Comfort during specific situation will be evaluated after 4 weeks of wearing the rigid socket and after 4 weeks of wearing the Access-Socket
  Score of the "Socket Comfort Score" scale. This scale is a visual analogic scale and ranges from 0 to 10. A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Loiret, PhD, Principal Investigator — Institut Régional de Médecine Physique et de Réadaptation de Nancy
Locations (4):
- France (4):
  - Hôpital d'Instruction des Armées (HIA) Percy, Clamart
  - Institut Régional de Médecine Physique et de Réadaptation de Nancy, Nancy
  - Centre d'Etudes et de Recherche sur l'Appareillage des Handicapés, Paris
  - Institution Nationale des Invalides, Paris

IPD SHARING:
Plan to Share IPD: No